CLINICAL TRIAL: NCT03457363
Title: Effect of the Adjunction of the Double Trunk Mask Above Standard Nasal Cannula
Brief Title: Double Trunk Mask and Standard Nasal Cannula During Acute Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratory of Movement, Condorcet, Tournai, Belgium (Other)
Responsible Party: Principal Investigator, frédéric Duprez, EPICURA ICU Hornu, Laboratory of Movement, Condorcet, Tournai, Belgium
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Duprezbruyneel
Record Dates: First submitted 2018-02-24; First posted 2018-03-07 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Hypoxia
Keywords: oxygen; nasal cannula; double trunk mask; hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Comparison of level oxygenation between classical oxygenation with nasal canulae with or without adjunctive of a double trunk mask
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double Trunk Mask (Experimental): DTM will be add above nasal cannula
  Interventions: Device: DTM will be add above NC
- Nasal Cannula Alone (Active Comparator): Patients receive oxygen only thought nasal Cannula
  Interventions: Device: DTM will be add above NC

INTERVENTIONS:
Device: DTM will be add above NC — After oxygenation by classical nasal cannula, the DTM will be place above NC

SUMMARY:
The objective of the study is to determine whether adjunctive mask of our design (Double Trunk Mask - DTM) has an effect on increasing arterial pressure in Oxygen (PaO2) diagnosed with severe hypoxia.

DETAILED DESCRIPTION:
This is a single-center, randomized, blind investigator, 2-way crossover study design. Enrolled participants had hypoxia being treated at Intensive Care Unit associated with a hospital in Hornu (Epicura).

The study consisted of two intervention periods separated by a washout period of 30 minutes.

The objective of the study is to determine whether adjunctive mask of our design (Double Trunk Mask - DTM) has an effect on increasing arterial pressure in Oxygen (PaO2) diagnosed with hypoxia.

The protocol and informed consent documents were reviewed and approved by a recognized ethics review board at the study facility. The study was performed in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Regardless of gender, at least 18 years of age and diagnosed with Hypoxia (PaO2/FiO2 < 380 mm Hg), dyspnea, respiratory rate (RR) ≥ 25 CPM, PaCO2 ≤ 45 mmHg, patient with an arterial catheter and without hemodynamic instability, Glasgow Coma Scale ≥ 12/15, written consent. Participants were also required to have a sufficient level of education to understand study procedures and be able to communicate with site personnel.

Exclusion Criteria:

* Patients were excluded if they Hypercapnia (> 45 mm Hg with respiratory acidosis), COPD, pulmonary fibrosis, hypoventilation obesity syndrome, arterial pressure < 60 mm Hg or treatment by epinephrine > to 0,1 gamma/kg/minute, deterioration of awareness (Glasgow scale < or = 12), acute confusional state.

Participants were randomized in a 1:1 ratio to receive either classical oxygenation with nasal cannula (NC) for 20 minutes or NC with an adjunctive of a Double Trunk Mask.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Oxygenation | 30 minutes
  we will observe effect of adjunction of a DTM on PaO2

SECONDARY OUTCOMES:
PaCO2 | 30 minutes
  we will observe the effect of the addition of the DTM on PaCO2

CONTACTS AND LOCATIONS:
Locations (1):
- Epicura, Hornu, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oude Nijhuis JC, Haane DY, Koehler PJ. A review of the current and potential oxygen delivery systems and techniques utilized in cluster headache attacks. Cephalalgia. 2016 Sep;36(10):970-9. doi: 10.1177/0333102415616878. Epub 2015 Nov 12. PMID 26566938
- [Background] Wettstein RB, Shelledy DC, Peters JI. Delivered oxygen concentrations using low-flow and high-flow nasal cannulas. Respir Care. 2005 May;50(5):604-9. PMID 15871753
- [Background] Tiep BL, Nicotra B, Carter R, Belman MJ, Mittman C. Evaluation of a low-flow oxygen-conserving nasal cannula. Am Rev Respir Dis. 1984 Sep;130(3):500-2. doi: 10.1164/arrd.1984.130.3.500. PMID 6476597

DOCUMENTS (3):
  • Study Protocol (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT03457363/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT03457363/SAP_001.pdf
  • Informed Consent Form (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT03457363/ICF_002.pdf